CLINICAL TRIAL: NCT00404768
Title: A Randomized, Double-blind, Placebo-controlled, Dose Ranging Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK221149A Administered Intravenously and to Investigate the Pharmacokinetics of GSK221149A Administered Orally to Healthy, Pregnant Females With Uncomplicated Pre-term Labor Between 300/7 and 356/7 Weeks' Gestation
Brief Title: The Safety, Tolerability And Metabolism Of GSK221149A, In Pregnant Women (30-36 Weeks), In Pre-Term Labor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OTA105256
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Obstetric Labour, Premature
Keywords: Premature Labor; Pre Term Labor; intravenous; fetal fibronectin
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — GSK221149A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Treatment (Experimental): GSK221149A
  Interventions: Drug: GSK221149A
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK221149A — 6mg/h and 12 mg/h
  Arms: Treatment
Drug: Placebo — Matched Placebo to Drug
  Arms: Placebo

SUMMARY:
Pre-Term Labor (prior to 37 weeks gestation) is the largest single cause of infant morbidity and mortality and is frequently associated with long-term disability. Oxytocin is a hormone produced by the body during labor. GSK221149A is an experimental drug that will be used to block the effects of oxytocin, and therefore pause or prevent contractions. In this study, patients with preterm labor will be given an intravenous infusion of GSK221149A over approximately 12 hours followed by an oral tablet in Parts A and B. In part C of this study, patients with preterm labor will be give an intravenous infusion of GSK221149A over approximately 48 hours. The use of a rescue tocolytic is allowed in the study.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, dose ranging study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK221149A administered intravenously and to investigate the pharmacokinetics of GSK221149A administered orally to healthy, pregnant females with uncomplicated pre-term labor between 300/7 and 356/7 weeks' gestation

ELIGIBILITY:
Inclusion criteria:

* Healthy pregnant females, 30 -36 weeks pregnant, without ruptured membranes
* 18-45 inclusive
* Symptoms of pre-term labor, (greater than or equal to 6 uterine contractions per hour, each of which at least 30 sec in duration, with cervical dilatation of less than or equal to 4 cm, (measured by tocodynamometry).

Exclusion criteria:

* Any clinically relevant abnormality identified on the screening examination or any other medical condition or circumstance making the patient (mother and/or fetus) unsuitable for participation in the study
* Any clinically relevant pre-existing or pregnancy-related co-morbid condition that may affect maternal pregnancy outcome or neonatal outcome (eg. hypertension, diabetes mellitus, bleeding/clotting diathesis)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2007-10-12 (Actual); Primary Completion 2011-07-07 (Actual); Study Completion 2011-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (29):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Colton, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Southern Pines, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Norfolk, Virginia
- GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina
- GSK Investigational Site, Sofia, Bulgaria
- GSK Investigational Site, Bogotá, Colombia
- France (5):
  - GSK Investigational Site, Clamart
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Poissy
  - GSK Investigational Site, Suresnes
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- GSK Investigational Site, San Juan, Puerto Rico
- GSK Investigational Site, Singapore, Singapore
- GSK Investigational Site, Seoul, South Korea
- Spain (4):
  - GSK Investigational Site, Barakaldo (Vizcaya)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia
- United Kingdom (3):
  - GSK Investigational Site, Warwick, Warwickshire
  - GSK Investigational Site, Coventry
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Jerry Snidow, Hugh Miller, Guillermo Valenzuela, Steve Thornton, Brendt Stier, Linda Clayton, Michael Fossler, Timothy Montague, Kathleen Beach, Pauline Williams. A Multicenter, Randomized, Double-blind Placebo-controlled Phase II Trial of Retosiban, a Selective Oxytocin Receptor Antagonist, for the Management of Preterm Labor. Am J Obstet Gynecol. 2013;2:S155.
- [Background] Thornton S, Valenzuela G, Baidoo C, Fossler MJ, Montague TH, Clayton L, Powell M, Snidow J, Stier B, Soergel D. Treatment of spontaneous preterm labour with retosiban: a phase II pilot dose-ranging study. Br J Clin Pharmacol. 2017 Oct;83(10):2283-2291. doi: 10.1111/bcp.13336. Epub 2017 Jul 11. PMID 28556962
- [Background] Thornton S, Miller H, Valenzuela G, Snidow J, Stier B, Fossler MJ, Montague TH, Powell M, Beach KJ. Treatment of spontaneous preterm labour with retosiban: a phase 2 proof-of-concept study. Br J Clin Pharmacol. 2015 Oct;80(4):740-9. doi: 10.1111/bcp.12646. Epub 2015 Jun 1. Erratum In: Br J Clin Pharmacol. 2015 Sep;80(3):609. doi: 10.1111/bcp.12694. PMID 25819462
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at multiple centers in the United States, United Kingdom, Singapore, France, Bulgaria, Spain, Argentina, South Korea, and Colombia from 03-December-2007 to 22-June-2011.
Groups:
- Part A/B: IV GSK221149A: Eligible participants received a single intravenous (IV) infusion of GSK221149A over 12 hours followed by a single oral dose of placebo tablets of strength 125 milligrams (mg) matched to GSK221149A. The GSK221149 loading dose and infusion rate were increased in a stepwise fashion every 3 hours to achieve plasma concentrations of 10, 30, 75, and 150 nanogram/milliliter (ng/mL).
- Part A/B: Oral GSK221149A: Eligible participants received placebo IV infusion over 12 hours followed by a single oral dose of GSK221149 125 mg tablets. The placebo loading dose and infusion rate were also increased every 3 hours in a stepwise fashion.
- Active (GSK221149A): Each participant received a loading dose of 6 mg GSK221149A over 5 minutes, followed by a constant IV infusion of 6 mg/h GSK221149A over 48 hours to reach a mean steady-state concentration (Css,ave) of 75 ng/mL.
- Placebo: Each participant received a loading dose of placebo over 5 minutes, followed by a constant IV infusion of placebo over 48 hours.
Period: Part A and B
Arm/Group | Part A/B: IV GSK221149A | Part A/B: Oral GSK221149A | Active (GSK221149A) | Placebo
Started | 20 | 9 | 0 | 0
Completed | 19 | 8 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawn due to labor progression | 1 | 0 | 0 | 0
Not completed — Withdrawn as delivery imminemnt | 0 | 1 | 0 | 0
Period: Part C
Arm/Group | Part A/B: IV GSK221149A | Part A/B: Oral GSK221149A | Active (GSK221149A) | Placebo
Started | 0 | 0 | 30 | 34
Completed | 0 | 0 | 22 | 20
Not Completed | 0 | 0 | 8 | 14
Not completed — Adverse Event | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Early withdrawal from study medication | 0 | 0 | 1 | 0
Not completed — Participant did not respond to therapy | 0 | 0 | 1 | 1
Not completed — Physician withdrew the study medication | 0 | 0 | 1 | 0
Not completed — Participant delivered baby | 0 | 0 | 0 | 1
Not completed — Unsatisfactory uterine response to IP | 0 | 0 | 0 | 1
Not completed — Active labor | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2
Not completed — Treatment failure | 0 | 0 | 0 | 1
Not completed — Investigator discretion | 0 | 0 | 0 | 1
Not completed — Researcher suspended study medication | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part A/B: IV GSK221149A: Eligible participants received a single IV infusion of GSK221149A over 12 hours followed by a single oral dose of placebo tablets of strength 125 mg matched to GSK221149A. The GSK221149 loading dose and infusion rate were increased in a stepwise fashion every 3 hours to achieve plasma concentrations of 10, 30, 75, and 150 ng/mL.
- Active (GSK221149A): Each participant received a loading dose of 6 mg GSK221149A over 5 minutes, followed by a constant IV infusion of 6 mg/h GSK221149A over 48 hours to reach a Css,ave of 75 ng/mL.
- Total: Total of all reporting groups
Arm/Group | Part A/B: IV GSK221149A | Active (GSK221149A) | Part A/B: Oral GSK221149A | Placebo | Total
Number analyzed (Participants) | 20 | 30 | 9 | 34 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.6 (4.97) | 25.2 (5.86) | 26.7 (5.66) | 27.8 (6.26) | 26.4 (5.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 30 | 9 | 34 | 93
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 2 | 3
  Asian | 2 | 2 | 1 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 2 | 7
  White | 17 | 23 | 8 | 24 | 72
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vital Sign Values of Potential Clinical Concern
Description: Vital signs included blood pressure (systolic and diastolic) and heart rate. Maternal blood pressure and heart rate were measured with the participant in the semi-supine position. Blood pressure was measured in millimeters of mercury (mmHg) and heart rate in beats per minute (bpm). Potential clinical concern range for systolic blood pressure: <85 and >160 mmHg, for diastolic: <45 and >100 mmHg and heart rate: <40 and >110 bpm. Only those parameters for which at least one value of potential clinical concern was reported are summarized. Number of participants with vital sign values of potential clinical concern are presented.
Time Frame: Up to Follow-up (Week 12)
Population: Safety Population which comprised of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part C: Active (GSK221149A): Each participant received a loading dose of 6 mg GSK221149A over 5 minutes, followed by a constant IV infusion of 6 mg/h GSK221149A over 48 hours to reach a Css,ave of 75 ng/mL.
- Part C: Placebo: Each participant received a loading dose of placebo over 5 minutes, followed by a constant IV infusion of placebo over 48 hours.
Arm/Group | Part A/B: IV GSK221149A | Part C: Active (GSK221149A) | Part A/B: Oral GSK221149A | Part C: Placebo
Number analyzed (Participants) | 20 | 30 | 9 | 34
Participants
  High heart rate | 2 | 4 | 0 | 3
  Low diastolic blood pressure | 1 | 4 | 0 | 4
  High diastolic blood pressure | 0 | 0 | 0 | 1
  Low systolic blood pressure | 0 | 3 | 0 | 4
  High systolic blood pressure | 1 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Values of Potential Clinical Concern
Description: All scheduled 12-lead ECGs were obtained after the participant was rested in the semi-supine position for approximately 15 minutes. Whenever 12-lead ECGs were performed at the same nominal time as a blood draw or blood pressure and pulse rate measurement, the 12-lead ECG were obtained first. ECGs were repeated or recorded in triplicate and the average value recorded at the investigators discretion. The potential clinical concern range for ECG parameters were: Absolute QT corrected (QTc) interval: >450 milliseconds (msec), Increase from Baseline (Day 0): QTc >60 msec, PR interval: <110 and >220 msec and QRS interval: <75 and >110 msec. All 12-lead ECGs obtained throughout the study day were evaluated for safety and were reviewed by the investigator or investigator designee. Number of participants with electrocardiogram values of potential clinical concern are presented.
Time Frame: Up to Follow-up (Week 12)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A/B: IV GSK221149A | Part C: Active (GSK221149A) | Part A/B: Oral GSK221149A | Part C: Placebo
Number analyzed (Participants) | 20 | 30 | 9 | 34
Participants | 13 | 15 | 8 | 9

3. Primary Outcome: Number of Participants With Clinical Chemistry and Hematology Parameter Values of Potential Clinical Concern
Description: Hematology parameters included complete blood count with red blood cell indices and white blood cell differential, platelet count, human immune deficiency virus, Hepatitis C antibody and Hepatitis B surface antigen. Clinical chemistry parameters included blood urea nitrogen (BUN), creatinine, glucose, sodium, potassium, phosphate, chloride, total CO2, calcium, aspartate amino transferase (AST), alanine amino transferase (ALT), gamma glutamyltransferase (GGT), alkaline phosphatase, total bilirubin, uric acid, albumin and total protein. Only those parameters for which at least one value of potential clinical concern was reported are summarized. Number of participants with clinical chemistry and hematology parameter values of potential clinical concern are presented.
Time Frame: Up to 24 hours post-treatment
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A/B: IV GSK221149A | Part C: Active (GSK221149A) | Part A/B: Oral GSK221149A | Part C: Placebo
Number analyzed (Participants) | 20 | 30 | 9 | 34
Participants | 10 | 22 | 7 | 28

4. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, is a congenital anomaly or birth defect. Any SAEs assessed as related to study participation (e.g. study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK product was recorded from the time a participant consents to participate in the study up to and including any follow-up contact.
Time Frame: Up to Follow-up (Week 12)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A/B: IV GSK221149A | Part C: Active (GSK221149A) | Part A/B: Oral GSK221149A | Part C: Placebo
Number analyzed (Participants) | 20 | 30 | 9 | 34
Participants
  AE | 11 | 14 | 2 | 17
  SAE | 1 | 2 | 0 | 2

5. Primary Outcome: Assessment of Amniotic Fluid Index (AFI)
Description: AFI is a quantitative estimate of amniotic fluid and an indicator of fetal well-being. AFI is the score (expressed in centimetes) given to the amount of amniotic fluid seen on ultrasonography of a pregnant uterus. An AFI between 8 to 18 is considered normal. An AFI < 5 to 6 is considered as oligohydramnios characterized by deficiency of amniotic fluid. An AFI > 18 to 24 is considered as polyhydramnios characterized by excess of amniotic fluid in the amniotic sac.
Time Frame: Up to 48 hours-post dose
Population: Pharmacodynamic Population which comprised of all participants who provided pharmacodynamic data. Data for only those participants available at the indicated time points were collected and analyzed. Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Part A/B: IV GSK221149A | Part C: Active (GSK221149A) | Part A/B: Oral GSK221149A | Part C: Placebo
Number analyzed (Participants) | 20 | 30 | 9 | 34
Score
  Pre-dose: number analyzed (Participants) | 20 | 29 | 8 | 34
  Pre-dose | 17.21 (6.213) | 11.86 (3.707) | 16.88 (4.295) | 13.34 (3.955)
  12 Hours: number analyzed (Participants) | 19 | 0 | 8 | 0
  12 Hours | 18.34 (5.208) |  | 12.98 (5.509) |
  24 Hours: number analyzed (Participants) | 0 | 23 | 0 | 22
  24 Hours |  | 13.15 (3.860) |  | 12.71 (4.662)
  48 Hours: number analyzed (Participants) | 0 | 25 | 0 | 21
  48 Hours |  | 13.38 (4.551) |  | 12.72 (4.379)

6. Primary Outcome: Number of Participants With 50% Reduction in Uterine Contractions Per Hour in Part A and B
Description: For uterine contraction assessment, an external tocodynamometer was fastened around the participant's abdomen. The number and duration of contraction was recorded at screening and up to 48 hours post-dose.The number of participants that achieve a reduction of at least 50% in uterine contractions with no cervical change within 6 hours and to maintain that reduction until 12 hours of therapy has been presented.
Time Frame: Up to 48 hours post-dose
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A/B: IV GSK221149A | Part A/B: Oral GSK221149A
Number analyzed (Participants) | 14 | 5
Participants | 9 | 1

7. Primary Outcome: Fetal Heart Rate Monitoring up to 48 Hours
Description: Fetal heart rate monitoring was incorporated to assess fetal tolerability. Fetal heart rate was monitored continuously at 2, 4, 6, 8, 12, 18, 24, 36 and up to 48 hours post-therapy. Mean fetal heart rate is presented. Data for only key-time points values have been presented.
Time Frame: Up to 48 hours post-dose
Population: Pharmacodynamic Population. Data for only those participants available at the indicated time points were collected and analyzed. Data points with null value for participants analyzed indicate data not collected for respective category and treatment arm.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A/B: IV GSK221149A | Part C: Active (GSK221149A) | Part A/B: Oral GSK221149A | Part C: Placebo
Number analyzed (Participants) | 20 | 30 | 9 | 34
Beats per minute
  Pre-dose | 140.0 (10.37) | 137.3 (7.77) | 134.8 (13.25) | 139.8 (8.49)
  2 Hours | 140.0 (9.41) | 138.4 (11.63) | 136.6 (10.27) | 137.4 (10.80)
  4 Hours: number analyzed (Participants) | 20 | 27 | 8 | 28
  4 Hours | 143.2 (11.44) | 133.0 (9.87) | 136.3 (11.88) | 138.3 (13.70)
  6 Hours: number analyzed (Participants) | 20 | 26 | 8 | 25
  6 Hours | 143.0 (10.37) | 133.0 (14.77) | 139.4 (14.00) | 137.1 (9.42)
  8 Hours: number analyzed (Participants) | 20 | 26 | 8 | 24
  8 Hours | 138.8 (10.51) | 133.2 (9.28) | 137.4 (11.69) | 134.1 (10.52)
  12 Hours: number analyzed (Participants) | 20 | 25 | 8 | 24
  12 Hours | 139.2 (9.95) | 135.7 (9.89) | 131.4 (9.97) | 135.4 (9.14)
  18 Hours: number analyzed (Participants) | 19 | 25 | 8 | 23
  18 Hours | 140.8 (9.27) | 138.7 (10.93) | 137.8 (11.42) | 135.4 (10.68)
  24 Hours: number analyzed (Participants) | 19 | 25 | 8 | 22
  24 Hours | 142.8 (12.17) | 139.6 (14.70) | 139.6 (10.47) | 135.2 (9.16)
  36 Hours: number analyzed (Participants) | 0 | 25 | 0 | 23
  36 Hours |  | 133.8 (10.88) |  | 137.4 (11.98)
  48 Hours: number analyzed (Participants) | 0 | 25 | 0 | 21
  48 Hours |  | 140.6 (13.64) |  | 140.5 (10.27)

8. Primary Outcome: Number of Participants Achieving Uterine Quiescence
Description: Uterine quiescence was defined as 4 contractions per/hour or less with no cervical change within the first 6 hours of therapy. Number of participants (from part A,B,C) achieving uterine Quiescence are presented.
Time Frame: Up to 48 hours post-dose
Population: Pharmacodynamic Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A/B: IV GSK221149A | Part C: Active (GSK221149A) | Part A/B: Oral GSK221149A | Part C: Placebo
Number analyzed (Participants) | 14 | 30 | 5 | 34
Participants | 9 | 18 | 2 | 13

9. Secondary Outcome: Number of Participants With Preterm Births in Part C
Description: Preterm is defined as babies born alive before 37 weeks of pregnancy are completed. There are sub-categories of preterm birth, based on gestational age: extremely preterm (<28 weeks) very preterm (28 to <32 weeks). Number of participants with preterm births are presented.
Time Frame: Up to 48 hours post-dose
Population: Pharmacodynamic Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Active (GSK221149A) | Part C: Placebo
Number analyzed (Participants) | 30 | 34
Participants | 5 | 16

10. Secondary Outcome: Neonatal Apgar Scores in Part A and B
Description: APGAR scores range from 0 to 2 for each condition (color, reflex response, muscle tone, respiration and heart rate) with a maximum final total score of 10. For heart rate: 0=no heart rate, 1=<100 bpm (baby not very responsive), 2=>100 bpm (baby vigorous); for respiration: 0=no breathing, 1= weak cry, 2=good, strong cry; for muscle tone: 0=limp, 1=some flexing of arms and legs, 2=active motion; for reflex response: 0=no response, grimace during stimulation, 2=grimace and cough or sneeze during stimulation; for color: 0=blue/pale, 1=good body color but blue hands and feet, 3=completely pink or good color. APGAR total score is the sum of sub-scores ranging from 0 to 10, where lower score indicates worst condition and higher score indicates best condition.
Time Frame: 1 minute and 5 minutes after birth
Population: Pharmacodynamic Population.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Part A/B: IV GSK221149A | Part A/B: Oral GSK221149A
Number analyzed (Participants) | 20 | 9
Scores on a Scale
  APGAR Five Minute Score | 8.8 (0.72) | 9.0 (0.00)
  APGAR One Minute Score | 7.7 (1.60) | 8.2 (0.67)

11. Secondary Outcome: Neonatal Weight Gain in Part A and B
Description: Neonatal safety was assessed through assessment of weight gain. Weight gain was measured at birth and follow-up (Week 12). Mean weight gain is presented.
Time Frame: At birth and Follow-up (Week 12)
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Part A/B: IV GSK221149A | Part A/B: Oral GSK221149A
Number analyzed (Participants) | 20 | 9
Grams
  At Birth | 3233.81 (478.8) | 3090.33 (643.2)
  At Follow-up | 4548.02 (809.1) | 4710.29 (818.0)

12. Secondary Outcome: Neonatal Head Circumference in Part A and B
Description: Neonatal safety was assessed through assessment of head circumference. Head circumference was measured at birth and follow-up (Week 12). Mean head circumference is presented.
Time Frame: At Birth and Follow-up (Week 12)
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Part A/B: IV GSK221149A | Part A/B: Oral GSK221149A
Number analyzed (Participants) | 20 | 9
Centimeters
  At Birth: number analyzed (Participants) | 19 | 9
  At Birth | 34.145 (1.6187) | 35.903 (7.7959)
  At Follow-up: number analyzed (Participants) | 19 | 9
  At Follow-up | 37.921 (5.1082) | 36.667 (1.5000)

13. Secondary Outcome: Neonatal Length Measured at 4-6 Weeks of Age in Part A and B
Description: Neonatal safety was assessed through assessment of neonatal length. Neonatal length was measured at birth and follow-up (approximately 4 to 6 weeks of age). Mean Neonatal length is presented.
Time Frame: At birth and follow-up (approximately 4 to 6 weeks of age)
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Part A/B: IV GSK221149A | Part A/B: Oral GSK221149A
Number analyzed (Participants) | 20 | 9
Centimeters
  At Birth | 50.3 (3.18) | 48.7 (3.64)
  At Follow-up: number analyzed (Participants) | 20 | 8
  At Follow-up | 54.6 (3.03) | 53.1 (3.04)

14. Secondary Outcome: Derived Plasma GSK221149 Pharmacokinetic Parameters- Area Under Concentration-time Curve From Time Zero to Infinity (AUC [0 to Infinity]) and Area Under Concentration-time Curve From Time Zero to Last Quantifiable Concentration (AUC [0 to Last])
Description: Blood samples (approximately 2mL) were collected for the PK measurement of plasma GSK221149 at pre-dose, 2, 4, 8, 12, 24 and 48 (just before infusion was stopped) hours after the start of the infusion.
Time Frame: Pre-dose, 2, 4, 8, 12, 24 and 48 (just before infusion was stopped) hours after the start of the infusion
Population: Safety Population. Only those participants who received oral GSK221149A 125 mg were assessed for PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | Part A/B: Oral GSK221149A
Number analyzed (Participants) | 8
Nanogram*hour per milliliter
  AUC infinity | 429.73 (40.1)
  AUC last | 419.09 (41.7)

15. Secondary Outcome: Derived Plasma GSK221149 Pharmacokinetic Parameters- Observed Elimination Half-life (T-half) and Time to Maximum Observed Drug Concentration (T-max)
Description: Blood samples (approximately 2 mL) were collected for the PK measurement of plasma GSK221149 at pre-dose, 2, 4, 8, 12, 24 and 48 (just before infusion was stopped) hours after the start of the infusion.
Time Frame: Pre-dose, 2, 4, 8, 12, 24 and 48 (just before infusion was stopped) hours after the start of the infusion
Population: Safety Population. Only those participants who received oral GSK221149A 125 mg were assessed for PK parameters
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A/B: Oral GSK221149A
Number analyzed (Participants) | 8
Hours
  T-half | 1.534 (0.6052)
  T-max | 1.713 (0.8286)

16. Secondary Outcome: Derived Plasma GSK221149 Pharmacokinetic Parameters- Maximum Plasma Concentration (Cmax)
Description: as for outcome 15
Time Frame: Pre-dose, 2, 4, 8, 12, 24 and 48 (just before infusion was stopped) hours after the start of the infusion
Population: Safety Population. Only those participants who received oral GSK221149A 125 mg were assessed for PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A/B: Oral GSK221149A
Number analyzed (Participants) | 8
Nanogram per milliliter | 126.93 (66.4)

17. Secondary Outcome: Neonatal Apgar Scores (at Birth) Measured at 4 to 12 Weeks Post Adjusted Gestational Age in Part C
Description: as for outcome 10
Time Frame: 1 minute and 5 minute after birth at 4 to 12 weeks post adjusted gestational age
Population: Pharmacodynamic Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part C: Active (GSK221149A) | Part C: Placebo
Number analyzed (Participants) | 30 | 34
Scores on a scale
  APGAR Five Minute Score | 9.0 (0.53) | 8.9 (0.34)
  APGAR One Minute Score | 8.3 (0.88) | 8.2 (0.77)

18. Secondary Outcome: Neonatal Weight Gain Measured at 4 to 12 Weeks Post Adjusted Gestational Age in Part C
Description: as for outcome 11
Time Frame: At birth and Follow-up (Week 12)
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Part C: Active (GSK221149A) | Part C: Placebo
Number analyzed (Participants) | 30 | 34
Grams
  At Birth | 3098.63 (512.644) | 2940.03 (584.950)
  At Follow-up: number analyzed (Participants) | 22 | 30
  At Follow-up | 3427.14 (635.5) | 3601.79 (659.479)

19. Secondary Outcome: Neonatal Head Circumference Measured at 4 to 12 Weeks Post Adjusted Gestational Age in Part C
Description: as for outcome 12
Time Frame: At Birth and Follow-up (Week 12)
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeteres
Arm/Group | Part C: Active (GSK221149A) | Part C: Placebo
Number analyzed (Participants) | 30 | 34
Centimeteres
  At Birth: number analyzed (Participants) | 27 | 34
  At Birth | 33.319 (1.7882) | 33.080 (1.6374)
  At Follow-up: number analyzed (Participants) | 21 | 27
  At Follow-up | 35.057 (1.7581) | 35.160 (1.7792)

20. Secondary Outcome: Neonatal Length Measured at 4 to 12 Weeks Post Adjusted Gestational Age in Part C
Description: Neonatal safety was assessed through assessment of neonatal length. Neonatal length was measured at birth and follow-up (Week 12). Mean neonatal length is presented.
Time Frame: At Birth and Follow-up (Week 12)
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Part C: Active (GSK221149A) | Part C: Placebo
Number analyzed (Participants) | 30 | 34
Centimeters
  At Birth: number analyzed (Participants) | 28 | 34
  At Birth | 47.8 (2.78) | 47.8 (3.39)
  At Follow-up: number analyzed (Participants) | 22 | 29
  At Follow-up | 50.6 (2.89) | 51.3 (3.30)

21. Secondary Outcome: Number of Participants Who Remained Undelivered Without Rescue Tocolytic Therapy After 48 Hours in Part C
Description: Tocolytics are medications used to suppress premature labor. They are given when delivery would result in premature birth. Number of participants who remained undelivered without rescue tocolytic therapy after 48 hours are presented.
Time Frame: 48 hours post-dose
Population: Pharmacodynamic Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Active (GSK221149A) | Part C: Placebo
Number analyzed (Participants) | 30 | 34
Participants | 30 | 34

22. Secondary Outcome: Percentage Reduction From Baseline in Number of Uterine Contractions [>30 Sec] Per Hour Within First 6 Hours of Therapy in Part C
Description: For uterine contraction assessment, an external tocodynamometer was fastened around the participant's abdomen. The number and duration of contraction was recorded at screening and up to 48 hours post-dose. Baseline was Day 0. Reduction from Baseline was calculated by subtracting Baseline values from post-Baseline values. Percentage reduction from Baseline in number of uterine contractions [>30 sec] per hour within first 6 hours of therapy are presented.
Time Frame: First 6 hours of therapy
Population: Pharmacodynamic Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part C: Active (GSK221149A) | Part C: Placebo
Number analyzed (Participants) | 30 | 34
Percent change
  1 Hour | -26.29 (45.406) | -19.03 (41.345)
  2 Hour | -36.65 (44.144) | -27.67 (58.181)
  3 Hour: number analyzed (Participants) | 29 | 31
  3 Hour | -49.14 (42.200) | -23.11 (68.820)
  4 Hour: number analyzed (Participants) | 27 | 29
  4 Hour | -62.06 (38.874) | -35.56 (69.171)
  5 Hour: number analyzed (Participants) | 26 | 26
  5 Hour | -59.20 (43.290) | -51.78 (49.544)
  6 Hour: number analyzed (Participants) | 26 | 24
  6 Hour | -65.32 (37.762) | -49.26 (47.871)

ADVERSE EVENTS:
Time Frame: Up to Follow-up (Week 12)
Description: Safety Population was used for adverse events assessment.
Arm/Group | Part A/B: IV GSK221149A | Part C: Active (GSK221149A) | Part A/B: Oral GSK221149A | Part C: Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/30 | 0/9 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/20 | 2/30 | 0/9 | 2/34
Other Adverse Events (participants affected / at risk) | 12/20 | 10/30 | 3/9 | 14/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A/B: IV GSK221149A (N=20) | Part C: Active (GSK221149A) (N=30) | Part A/B: Oral GSK221149A (N=9) | Part C: Placebo (N=34)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Amniotic fluid volume decreased (Investigations) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cerebral atrophy congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A/B: IV GSK221149A (N=20) | Part C: Active (GSK221149A) (N=30) | Part A/B: Oral GSK221149A (N=9) | Part C: Placebo (N=34)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Labour pain (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Postpartum depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Developmental delay (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macrocephaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neonatal pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment neonatal (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteral disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection neonatal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.